CLINICAL TRIAL: NCT01017419
Title: Orientation for Hearing Aid Users: Information Retention
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Deborah Viviane Ferrari, Faculdade de Odontologia de Bauru - Universidade de São Paulo
Other Study IDs: 3
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Hearing Loss
Keywords: hearing aids; counseling
MeSH Terms: conditions — Hearing Loss | interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Audiology counseling
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Informational Counseling provided after hearing aid fitting

SUMMARY:
Aim: To verify how much of the orientation provided at diagnosis and hearing aid fitting are retained by new hearing aid users and analyze whether age, degree of hearing loss, academic and socio-economics status have an influence on this

DETAILED DESCRIPTION:
Introduction: The understanding and retention of orientations provided by the health professional increases patient's satisfaction and compliance to treatment and reduces treatment duration and costs. Aim: To verify how much of the orientation provided at diagnosis and hearing aid fitting are retained by new hearing aid users and analyze whether age, degree of hearing loss, academic and socio-economics status have an influence on this. Methods: Participated in this study 30 adults (18 female and 12 male) with age varying from 18 to 88 years, with post lingual uni or bilateral hearing loss of various degrees and types. Orientations were offered at the time of diagnosis and hearing aid fitting. At the first follow up visit patients were interviewed regarding their hearing loss' characteristics as well as hearing aid care and use (probed recall task). It was also evaluated how participants manipulated their devices. A protocol was used to score participant's responses. Results: on average participants could retain 31,6% and 83,6% of the orientation provided regarding their hearing loss and hearing aid care and use. There was a negative correlation between age and amount of information retained. There was no influence of degree of hearing loss, academic and socio-economic statues. Conclusion: The hearing impaired patients have difficulty to recall orientation provided therefore the use of facilitation strategies to information retained is necessary.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* sensorineural hearing loss, hearing aid candidate

Exclusion Criteria:

* severe dexterity or visual problems. Cognitive or memory disorders

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adults (18 female and 12 male) with age varying from 18 to 88 years, with post lingual uni or bilateral hearing loss of various degrees and types.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah V Ferrari, Doctor, Principal Investigator — University of Sao Paulo
Locations (1):
- Hrac - Usp, Bauru, São Paulo, Brazil